CLINICAL TRIAL: NCT02723643
Title: Initial Investigation on Potential Associated Factors of Uncontrolled Hypertension in Outpatient Department: A Prospective Registry Study
Brief Title: Potential Associated Factors of Uncontrolled Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GDREC 2015373H
Record Dates: First submitted 2016-03-18; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension,Essential
Keywords: Hypertension; Essential hypertension; Blood pressure; Cardiovascular diseases
MeSH Terms: conditions — Essential Hypertension; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Venous blood will be sampled for further DNA assessment after informed consent is obtained

SUMMARY:
The incidence and prevalence of hypertension is increasing while the controlled rate is extremely low in China. A substantial percentage of participants with uncontrolled hypertension are correctable if potential associated factors are identified and corrected. Therefore, it is clinically relevant to investigate and identify these potential associated factors of uncontrolled hypertension so as to increase controlled rate and reduce hypertension-associated health and economic burdens in the future. Investigators plan to conduct a prospective registry study in a single-center to initially investigate the potential associated factors of uncontrolled hypertension in cardiovascular outpatient department. Furthermore, investigators plan to evaluate the effects of potential associated factors correction on hypertension controlled rate and cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinic systolic and/or diastolic blood pressure above 140 and/or 90 mm Hg treating with 3 different classes of anti-hypertensive drugs (not necessarily including diuretic).

Exclusion Criteria:

* Known secondary hypertension,
* Pregnant women,
* Chronic kidney disease (CKD) 3 or higher,
* Has a history of connective tissue diseases,
* Has a history of any type of cancer,
* Cognitive disorder which could not finish home blood pressure monitoring,
* Has a history of coronary heart disease,ischemic stroke,transient ischemic attack or heart failure.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient populations with clinic systolic and/or diastolic blood pressure above 140 and/or 90 mm Hg treating with 3 different classes of anti-hypertensive drugs (not necessarily including diuretic).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Hypertension controlled rate in participants after potential associated factors are corrected | Up to 1 month
  Participants with uncontrolled hypertension (SBP and/or DBP >=140 and/or 90 mm Hg) treating with 3 or more anti-hypertensive drugs (not necessarily including diuretic) in outpatient department will under assessment of hypertension controlled rate 1 month later after initial investigation of potential associated factors. Based on these findings, investigators will give instructions to participants how to correct those potential associated factors and follow-up participants via telephone or outpatient visit 1 month later to assess whether these corrections could help increase hypertension controlled rate. Participants will be required to record home blood pressure measurements every day, and average home SBP and DBP will be calculated 1 month later. If average home SBP/DBP < 135/85 mm Hg then participants will be considered as controlled-case, otherwise uncontrolled case.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Cardiovascular Institute,Guangdong General Hospital, Guangzhou, Guangdong, China